CLINICAL TRIAL: NCT03923452
Title: Mindfulness Training for Low-Income Older Adult Canadian Immigrants
Brief Title: Mindfulness Training for Older Adult Canadian Immigrants
Acronym: MTCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Toronto Metropolitan University (Other)
Responsible Party: Principal Investigator, Alexandra J. Fiocco, PhD, Associate Professor, Toronto Metropolitan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AFiocco
Record Dates: First submitted 2019-04-18; First posted 2019-04-22 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2024-04

CONDITIONS: Stress
Keywords: mindfulness; immigrant; stress; wellbeing
MeSH Terms: interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Intervention Model Description: Randomized block design: 25 randomized to experimental group; 25 randomized to control group in blocks of 8
Who Masked: Outcomes Assessor
Masking Description: Researcher who engage in pre-post testing assessment will be blinded to participant allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MBSR: Mindfulness-based stress reduction (Experimental): Participants will be exposed to the 9-week MBSR program, facilitated by a trained MBSR facilitator. Due to COVID-19, the program will be held virtually.
  Interventions: Behavioral: Mindfulness-based Stress Reduction
- WLC: Wait list Control (No Intervention): Participants will be asked to log their self-care activities every week.

INTERVENTIONS:
Behavioral: Mindfulness-based Stress Reduction — Mindfulness-based stress reduction is a manualized mindfulness training protocol that has been researched for over 20 years. The original protocol will be used, with the exception of the prescribed home practice duration (i.e. 30 mins of practice). Rather, the program will be modified to set up participants for success by providing them with instruction to "build" on their meditation practice, beginning with 8 minutes a day.
  Arms: MBSR: Mindfulness-based stress reduction

SUMMARY:
This study will evaluate whether mindfulness-based stress reduction (MBSR) is a viable community program for enhancing wellbeing among older adult immigrants from low income neighborhoods. Half of the sample will be randomized to receive the 9-week mindfulness program and the other half will be randomized to a wait list control condition. Primary outcomes of interest will include perceived stress and self-report depressive symptoms. Secondary outcomes will include trait mindfulness and self-care, self-compassion, emotion regulations, and attentional skills. Participants will also be invited to engage in a 30-minute interview to discuss their lived experience as an immigrant in Canada and their experience in the MBSR program. Due to COVID-19, all sessions will be held virtually.

DETAILED DESCRIPTION:
Adults aged 65 years and older are the fastest growing segment of the Canadian population. In the 2006 Census, 43% of older adults in Ontario identified as being a Canadian immigrant, a statistic which continues to grow in the context of an aging population. Aging is commonly associated with declines in physical and cognitive capacity, which is significantly accelerated by chronic perceived stress. Lower income older adults are particularly vulnerable to accelerated aging and disease onset due to the stress of economic insecurity. In 2012, the highest low-income rates in Canada were reported among immigrants 65 years of age and older. Accordingly, it is important to investigate programs that can support the wellbeing of aging Canadian immigrants.

The principal investigator (PI) and her research team will conduct a one-factor between-subjects design with two conditions - a mindfulness-based intervention and a waitlist control - to examine the benefits of mindfulness training on indices of wellbeing, including perceived stress, depressive symptoms, emotion regulation, self-compassion and self care. It is hypothesized that mindfulness training will enhance indices of wellbeing compared to a wait-list control. Employing a mixed-methods approach, participants will also engage in a qualitative interviews to provide insight into the lived experience and how mindfulness may serve Canadian immigrants.

ELIGIBILITY:
Inclusion Criteria:

* 60+ years of age; Canadian immigrant; low socioeconomic status; immigrated to Canada within last 15 years; reports experiencing stress in their daily life.

Exclusion Criteria:

* existing contemplative practice; currently enrolled in a research study; non-fluency in English; neurological disorder that prevents participation in the 9-week program or testing procedures; plans to vacation during the study period/unable to attend 9 program sessions and 2 testing sessions; existing substance abuse (last 6 months); psychiatric disorder that may prevent participation in 9-week program or testing procedure.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-06-30 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Perceived Stress Scale (PSS) | 2 days (pre-post testing)
  the PSS is a 14-item questionnaire that measures general perceived stress. Total Scores range from 0-56, with higher scores denoting greater perceived stress.
Center for epidemiological studies - depression (CES-D) | 2 days (pre-post testing)
  The CES-D is a self-report measure of depressive symptoms. Total score ranges from 0-60, with greater scores denoting greater endorsement of depressive symptoms.

SECONDARY OUTCOMES:
Five Facet Mindfulness Questionnaire (FFMQ) | 2 days (pre-post testing)
  The FFMQ is a 33-item self-report measure, that measures mindfulness characteristics including the ability to observe, describe, act with awareness, non-judging, and non-reacting. ". Subscale scores range from 8 to 40 for the observing, describing, acting with awareness, and non-judging facets, or 7 to 35 for the non-reacting facet, resulting in an overall FFMQ score range of 39 to 195. Higher scores indicate greater levels of TM.

OTHER OUTCOMES:
Difficulties in Emotion Regulation Scale (DERS-16) | 2 days (pre-post testing)
  A 16-item Likert-type scale that measure the propensity for emotion regulation. Higher scores indicate greater emotion regulation.
Mindful Self-Care Scale- SHORT (MSCS) | 2 days (pre-post testing)
  The Mindful Self-Care Scale- SHORT (MSCS, 2016) is a 33-item scale that measures the self-reported frequency of behaviors that measure self-care behavior.The scale addresses 6 domains of self-care: physical care, supportive relationships, mindful awareness, self-compassion and purpose, mindful relaxation, and supportive structure.
Stroop Task | 2 days (pre-post testing)
  A 15-minute computer-based task that measures attention and inhibition.
Self-Compassion Scale (SCS) | 2 days (pre-post testing)
  A 26-item Likert-type scale (Almost Never to Almost Always) that measures self-compassion. Greater scores indicate greater self-compassion.
Brief Resilience Scale (BRS) | 2 days (pre-post testing)
  A 6-item Likert-type scale (Strongly Disagree to Strongly Agree) that measures resilience when faced with challenge and set-backs. Higher scores indicate greater resilience.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra J Fiocco, PhD, Principal Investigator — Toronto Metropolitan University
Locations (1):
- Toronto Metropolitan University (formerly Ryerson University), Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
de-identified quantitative data will be posted on an open science framework when published in an open access journal. Data will also be made available upon request under ethical guidance.